CLINICAL TRIAL: NCT06796608
Title: Technology-Supported Behavioral Activation to Optimize Day-to-Day Quality of Life With Advanced Cancer
Brief Title: Behavioral Activation-Led Activity Engagement for Cancer Empowerment
Acronym: BALANCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Carissa Low, Associate Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY24010177
Record Dates: First submitted 2024-12-18; First posted 2025-01-28 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Advanced Cancer; Cancer
Keywords: behavioral activation; quality of life
MeSH Terms: conditions — Neoplasms | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Activity tracking via smartphone app (Experimental): Participants will rate their day and indicate activities they did that day via the smartphone once each evening for the first four weeks. After four weeks, they will complete a mid-study data review session with a study team member about the activities, behaviors, and experiences they believe are most strongly related to their day-to-day quality of life. For the last 4 weeks of the study, they will select at least 4 behaviors or activities to increase. Participants will fill out morning surveys to plan an activity, receive daily reminders through the BALANCE app to support behavior change, and complete evening surveys to report daily quality of life and indicate completed activities.
  Interventions: Behavioral: Behavioral Activation

INTERVENTIONS:
Behavioral: Behavioral Activation — Behavioral activation is an evidence-based intervention based on the idea that depression leads to withdrawal from rewarding activities, which sustains or exacerbates depression, and breaks this cycle by increasing the frequency with which people engage in rewarding activities regardless of their motivation. Like those with depression, people living with advanced cancer may reduce or stop participation in meaningful life activities resulting in decreased positive emotion and worse quality of life. The goal of this intervention is to adapt and test a fully remote technology-supported behavioral activation intervention aimed at supporting patients with advanced cancer to optimize the quality of their remaining years of life.
  Other Names: Behavioral Intervention; Behavior Modification; Behavior or Life Style Modifications

SUMMARY:
The goal of this study is to learn if behavioral activation can improve daily quality of life for patients with advanced cancer. The main questions it aims to answer are:

* Can behavioral activation be adapted to help patients living with advanced cancer optimize their daily quality of life?
* Can behavioral activation be delivered primarily via smartphone?

Participants will:

* Complete a demographic questionnaire at the beginning of the study and quality-of-life and activity questionnaires at the beginning, midpoint, and end of study. Complete nightly surveys about daily quality of life, mood, activities, and experiences.
* Wear a Fitbit activity tracker for 8 weeks.
* After the first four weeks, they will complete a session with a member of our team about their day-to-day activities, behaviors, and experiences. They will select at least 4 activities/behaviors to increase over the next portion of the study.
* Incorporate personalized meaningful activities into daily life
* At the end of approximately eight weeks, (four weeks after the session with a study team member), they will complete a semi-structured interview.

DETAILED DESCRIPTION:
Participants (n=25) will be recruited from UPMC Hillman clinics.

Part 1 (Consent and Baseline data collection from weeks 1 to 4):

If eligible patients consent to participate, they will complete online baseline questionnaires. Participant's medical records will be reviewed to extract demographic information and clinical covariates, including information about their cancer, its treatment, biological variables such as sex and age, clinical variables such as comorbidities, surgeries and hospitalizations, medications, and other markers of health care utilization (e.g., emergency department visits). Once extracted, these values will be linked only to their study ID number.

At the initial visit (either in-person or online, 20-30 minutes), participants will also be oriented to the ecological momentary assessment procedures to assess self-reported daily quality of life and mood, activities, and experiences. Participants will install the BALANCE Android or iOS application on their smartphones. The participant ID will be entered into the app upon initial log in and will be saved locally on the device. Participants will have the opportunity to add additional activities to track for 2 days before the 4 weeks of Part 1 of the study begins. When participants receive the survey notification, it will open the application and they can proceed to take the survey in the BALANCE app on their smartphone. Participants will be asked to complete the EMA questions once each evening (approximately 5 minutes). Participants will be able to use the BALANCE app to access visualizations of their past survey responses and quality of life ratings along with activity and sleep data.

Participants will also be asked to wear a Fitbit device (Fitbit Inspire 3 or similar) for the duration of the study and to install the Fitbit app on their smartphone. The Fitbit is a wristwatch-sized waterproof device that assesses heart and breathing rates, physical activity, and sleep, skin temperature, and oxygen levels and wirelessly transmits data to the server. If they already own a Fitbit device, we will request access to their Fitbit data for the duration of their study participation.

Mid-Study Data Review (mid-study data review session following first 4 weeks of the study):

Participants will complete a mid-study data review session (in person or remotely, 20-30 minutes) with a member of our team during which they will be asked which activities, behaviors, and experiences they believe to be the most strongly related to their day-to-day quality of life. They will also be provided with the results of personalized analyses visualizing the factors most strongly correlated with their quality of life ratings over the past four weeks. Based on their own reflections and these personalized analyses, they will be asked to select at least 4 behaviors or activities to increase over the next four weeks. Participants will also complete a midpoint questionnaire at this time.

Part 2 (Data-based intervention from mid-study data review session to approximately 8 weeks):

For the second four weeks of the study, starting after the mid-study data review session with a study team member, participants will complete a morning survey to make a plan for behavior change, receive daily reminders to complete their planned activities through the BALANCE Android or iOS application on their smartphones, and will complete an evening survey to report their daily quality of life and indicate completed activities (both < 5 minutes) each day. Participants will also collect Fitbit data during the same period. At the end of this second 4-week period, we will invite participants for a 1-on-1 in-person or online semi-structured interview (20-30 minutes) to provide feedback. In addition, we will assist participants in removing the BALANCE app from their phones. Participants will also complete an end of study questionnaire at this time.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with Stage IV cancer and receiving ongoing treatment at a UPMC Hillman Cancer Center clinic
* owns and uses a smartphone capable of running study applications

Exclusion Criteria:

* Unable to read, write, or communicate in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2025-01-28 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Acceptability | At end of intervention at approximately 8 weeks
  Post-intervention semi-structured interviews will be conducted to gather participant feedback and assess acceptability of the program
Acceptability | At the end of intervention at approximately 8 weeks
  System Usability Scale (SUS). For odd items, subtract one from the user response. For even-numbered items, subtract the user responses from 5.
  This scales all values from 0 to 4 (with four being the most positive response).
  Add up the converted responses for each user and multiply that total by 2.5. Possible range of scores is 0 to 100 representing a composite measure of the overall usability of the system being studied.
Feasibility | From enrollment to the end of intervention at approximately 8 weeks
  accrual rate (number of participants that enroll out of number of participants approached)
Feasibility | From enrollment to the end of intervention at approximately 8 weeks
  completion rate (number of participants that complete the study)
Feasibility | From enrollment to the end of intervention at approximately 8 weeks
  engagement (how many days within the study the participants engaged with the app and had Fitbit data)

SECONDARY OUTCOMES:
Daily ratings | Change from baseline to the end of intervention at approximately 8 weeks
  Participants' average daily quality of life rating from 0 to 10 (with higher values indicating better days)
Quality of Life | Change from baseline to the end of intervention at approximately 8 weeks
  Patient-Reported Outcome Measurement Information System (PROMIS) 29+2 is used to evaluate general health-related quality of life. The seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance) have four items per domain and use a 5-point Likert response scale. Possible range of scores for these 7 domains is 4 to 20. The pain intensity item uses a numeric rating scale (0 [no pain] to 10 [worst pain imaginable]). The sum of raw scores for each domain is converted into a standardized T-score using a publicly available conversion table or an online scoring service. Higher scores represent worse symptoms for symptom-oriented domains (anxiety, depression, fatigue, pain intensity, pain interference, and sleep disturbance) and better health outcomes for function-oriented domains (physical functioning and ability to participate in social roles and activities).
Depressive symptoms | Change from baseline to the end of intervention at approximately 8 weeks
  Center for Epidemiologic Studies Depression Scale (CES-D Scale). Possible range of scores is 0 to 60, with the higher scores indicating the presence of more symptomatology.

OTHER OUTCOMES:
Restorative Activities | Change from baseline to the end of intervention at approximately 8 weeks
  Pittsburgh Enjoyable Activities Test (PEAT). Participants are asked how often they have participated in a number of leisure activities during the past month. Possible range of scores is 0 to 40. Higher PEAT scores indicate more time spent doing leisure activities.
Objective physical activity | Change from baseline to the end of intervention at approximately 8 weeks
  A Bluetooth enabled activity monitor worn throughout the study will estimate number of steps/day.
Activity disruption | Change from baseline to the end of intervention at approximately 8 weeks
  Sickness Impact Profile short form (6 items) is used to assess a person's perception of their health status with respect to their disease impact. Possible range of scores is 0 (0%) to 6 (100%). Higher scores represent poor health status or a major impact of illness on behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Carissa A Low, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Preliminary IPD data from this pilot study will not be shared